CLINICAL TRIAL: NCT02695576
Title: Lumbar Fusion or Non-operative Care for Treatment of Presumed Discogenic Pain: A Randomized Study
Brief Title: Lumbar Fusion or Non-operative Care for Treatment of Presumed Discogenic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spinal Surgery Clinic, Strängnäs (Other)
Responsible Party: Principal Investigator, Bo Nyström, MD, PhD, Spinal Surgery Clinic, Strängnäs
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SpinalSC
Record Dates: First submitted 2016-02-02; First posted 2016-03-01 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Physical Therapy Modalities; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgery (Experimental): Lumbar fusion surgery Physiotherapy Cognitive behavioral therapy
  Interventions: Procedure: Lumbar Fusion Surgery; Other: Physiotherapy; Other: Cognitive behavioral therapy
- Non-surgery (Active Comparator): Physiotherapy Cognitive behavioral therapy
  Interventions: Other: Physiotherapy; Other: Cognitive behavioral therapy

INTERVENTIONS:
Procedure: Lumbar Fusion Surgery — Interbody fusion with fixation
  Arms: Surgery
Other: Physiotherapy — Examination by physiotherapist, motivation of the patient, training in body awareness, physical activity/Qigong, training in water, outdoor pole work, circle training, stabilization training, massage, stretching, lessons and practice in ergonomics.
Other: Cognitive behavioral therapy — Individual and group lessons performed by psychologists.

SUMMARY:
Title and abstract

1 a. Title: Lumbar fusion or non-operative care for treatment of presumed discogenic pain.

A randomized study.

1 b. Structured summary:

Authors: B. Nyström, B. Schillberg, E. Svensson, T. Stiles.

Corresponding author: Bo Nyström, Clinic of Spinal Surgery, Strängnäs, Sweden. e-mail address: pgbo.nystrom@gmail.com

Background: At present there is no clear evidence that surgical treatment by fusion operation is more advisable than non-surgical treatment in patients suffering from unspecific chronic low back pain (CLBP). By personal experience a subgroup among the CLBP patients is selected, possibly representing patients with pain from a motion segment/disc, thus making patient selection more specified. Furthermore, selection of level to fuse based on radiological findings has not been found reliable. Therefore a mechanical provocation test has been developed at the clinic. The aim of this randomized study was to compare the outcomes in pain and pain related functions perceived by this specific subgroup of CLBP patients following fusion surgery with those following non-surgical treatment.

Methods: Patients with a specified symptomatology and specified clinical signs at examination were recruited and randomized to either type of treatment, non-surgical (NS) including cognitive-behavioral therapy and physiotherapy (37 pat.) or surgical (S), including the same cognitive-behavioral therapy and physiotherapy as in the NS group plus fusion surgery (37 pat.). All patients were thoroughly investigated before start of the study and at follow-up one year after treatment. The outcomes perceived by the patients were assessed on the validated questionnaires Oswestry Disability Index (ODI), Roland-Morris, Balanced Inventory for Spinal Disorders (BIS), Short-Form-36 (SF-36) and Euro-Quol (EQ-5D).

DETAILED DESCRIPTION:
1. a. Title: Lumbar fusion or non-operative care for treatment of presumed discogenic pain.

   A randomized study.

   Introduction

   Background and objectives:
2. a. Only two out of five existing randomized studies comparing results from fusion surgery for chronic low back pain (CLBP) with results from conservative treatment have reported the results from surgery to be better. Systematic review of these trials also found methodological concerns. At present, therefore, there is no clear evidence that surgical treatment is more advisable than non-surgical treatment in patients suffering from unspecific CLBP.

2 b. The investigators hypothesis is that a/ there exists a specific identifiable subgroup of patients within the CLBP group in whom the pain emanates from the disc, and that b/ patients in this subgroup may be selected based on thorough symptom analysis, and c/ that the actual disc may be localized, not by radiological methods or discography, but by mechanical testing procedures, making pain reduction possible by a fusion operation at that level.

Methods

Trial design:

3 a. A RCT with parallel group design with pre- and post-treatment data.

3 b. No changes were made after trial commencement.

Participants

4 a. Inclusion criteria: 18 to 65 years, with pronounced low back pain for at least one year and having tried ordinary physical therapy without improvement and being on sick leave at least 50 %. They should not have had any prior fusion operation but may have had surgery for e.g. a disc herniation.

4 b. Eligible outpatients at the Clinic of Spinal Surgery, Strängnäs, Sweden, were informed about the study and those who consented to participate were included, the other received ordinary treatment outside the study.

Data were collected at the Clinic of Spinal Surgery, Strängnäs, Sweden. Interventions

5. A percutaneous mechanical provocation test was developed to obtain information regarding a possibly painful segment. Local disc injections were also performed to analyse the pain response at needle contact with the disc, at injection into the disc with saline or local anaesthetics blind for the patients and also the pain situation following local anaestetics into the disc, discoblock.

Further, an open mechanical provocation test was developed to analyse the location of a possibly painful disc. Operation by posterior lumbar interbody fusion was performed using microsurgical technique and autologous bone. Internal fixation was used.

Patients in both groups, the surgical (S) and the non-surgical (NS) group, were all treated by formal physiotherapy at a five days stay at the Clinic and instructed to continue their training at home according to the lines given at the Clinic. Patients in both groups were similarly treated individually by cognitive-behavior therapy at seven occasions.

Outcomes

6 a. The primary outcome was back pain, assessed by the patients on the BIS and on a VAS before treatment and at follow-up one year after treatment as well as the perceived change in pain.

Secondary outcomes were pain related functions assessed on the ODI, the Roland-Morris, and the BIS questionnaires. Health related quality of life was also assessed as a secondary outcome measure, by using the SF-36 and EQ-5D questionnaires.

6 b. No changes in trial outcomes were made during the study.

Sample size

7a. The sample size calculation was performed before study start by the statistician (ES). It was based on previous knowledge of outcomes from a Swedish cross-sectional study (surgery vs physiotherapy) in which the proportions patients with improvement were 63% and 29%, respectively. Assuming similar results of improvements a total sample size of 66 (33+33) will detect such a difference with the statistical power of 80%.

7 b. Interim analysis did not occur.

Randomization. Sequence generation.

8 a and b. A randomization scheme balanced for female/male, as well as for surgery/non-surgery patients was performed by using random permuted blocks of 20 (10 females and 10 male) patients in order to reduce predictability. The permutation blocks were randomly chosen. Two sets of closed envelopes in numbered orders, one set for males and one for females, with either message "operate" or "do not operate" were delivered to the clinic by the statistician not involved in the treatment of the patients.

Allocation concealment mechanism

9. The patients were consecutively included in the study according to the randomization envelopes.

Implementation

10. A statistician not involved in the treatment of the patients generated the random allocation sequence. The surgeon enrolled the participants and an anaesthesiology nurse at the clinic performed the practical assignment, i.e. opened the closed envelopes in consecutive order.

Blinding

11 a. In accordance with the treatment alternatives the participants and the care givers could not be blinded to group assignment.

11 b. Patients in both groups, the surgical and the non-surgical, received equal cognitive-behavioral treatment and physiotherapy. Besides, patients in the surgical group were operated by spinal fusion.

Statistical methods

12 a and b. The outcome variables are assessed on rating scales that generate ordered categorical data. Characteristic features are the ordered structure with lack of information regarding size and inter-categorical distances. Non-parametric rank-based statistical methods that take account of these limited mathematical properties of ordered categorical data have been used for description and analysis. Frequency distribution, proportions, bar charts, median and quartiles are used for statistical description of cross-sectional data. Statistical analysis of difference in outcomes assessed by transitional scales in the BIS by the two groups of patients was performed by the Wilcoxon-Mann-Whitney test. Statistical evaluation of change in the paired assessments made before treatment and on the follow-up occasion was made by a statistical approach developed for paired ordinal data that provides measures of systematic change in common for the group and additional measure of individual variability. The measures and the 95% confidence intervals of systematic change in position (RP), and in concentration (RC), and the measure of individual variability (RV) will be calculated as well as the differences in these measures between the two treatment groups. This approach has been found to have a high power of detecting differences in small samples.

Results

13. All patients in the surgical as well in the non-surgical group received the allocated treatment. All patients in both groups were seen at follow-up.

Recruitment

14 a. Recruitment started July 4, 2007 and ended when the last patient was included in the study at March 28, 2011.

The follow-up took place from Oct. 21, 2008 to June 27, 2012.

14 b. The trial was performed as planned.

Numbers analysed

16. The analysis was carried out on the complete groups of 37 patients in each group and no missing patients.

Outcome and estimations

17 a and b. The material is not fully analysed yet.

Ancillary analysis

18. None.

Harms

19. There were no surgical complications, no neurological deterioration and no device failures. Five of the 37 patients in group S had defect bone healing and were re-operated by anterior fusion at the same level, one patient had anterior fusion at a new level and in 3 patients the fixation screws were extracted due to local pain.

Comment

Limitations:

20. There was a rather small sample size because of difficulties in recruiting eligible patients, but a good research team and the choice of appropriate statistical analysis shows the power of this study.

Generalizability

21. The investigators regard the results generalizable, provided that the patients and the level to fuse being selected according to the same criteria as in the present study.

Interpretation

22. Based on the results from existing randomized studies comparing fusion surgery with conservative treatment in patients suffering from CLBP it has not been evident that surgery is advisable. However, in previous studies the symptoms of the patients selected has been described simply as "chronic low back pain". The patients in the investigators study were selected based on a more specific symptom analysis. Furthermore, in previous studies the level to fuse has been chosen based on radiological findings whereas a mechanical provocation tests is used in the present study. Two of the previous studies stated the importance of cognitive-behavioral therapy in CLBP patients, resulting in equally good results as following fusion surgery. To study the specific effect of surgery, therefore, both groups in the investigators study received quite the same treatment with cognitive-behavioral therapy and physiotherapy, the difference between the two groups being that one group also received surgery.

Other information

Registration:

23. The study protocol was approved by the Regional Ethics Committee, Stockholm (reference number 2007/598-31/4). In accordance with the Declaration of Helsinki, all patients were thoroughly informed concerning all parts of the study, both verbally and in written text, and gave their written informed consent.

24. The full trail protocol can be accessed via Bo Nyström, Clinic of Spinal Surgery, Strängnäs, Sweden.

25. The study had no funding support.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain
* Clinical diagnosis
* No radiological correlates

Exclusion Criteria:

* No previous fusion operation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2007-07 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Low back pain assessed with Visual Analog Scale | One year
  Visual Analog Scale for Pain
Low back pain assessed with Balanced Inventory for Spinal Disorders (BIS) | One year
  Balanced Inventory for Spinal Disorders (BIS)
Low back pain assessed with Oswestry Disability Index (ODI) | One year
  Oswestry Disability Index (ODI)
Low back pain assessed with Short-Form-36 (SF-36) | One year
  Short-Form-36 (SF-36)

SECONDARY OUTCOMES:
Pain related functions assessed with Roland-Morris questionnaire | One year
  Roland-Morris questionnaire
Pain related functions assessed with European Quality-of-Life Scale (EQ-5D) | One year
  European Quality-of-Life Scale (EQ-5D)
Pain related functions assessed with Balanced Inventory for Spinal Disorders questionnaire (BIS) | One year
  Balanced Inventory for Spinal Disorders questionnaire (BIS)
Pain related functions assessed with Short-Form-36 questionnaire (SF-36) | One year
  Short-Form-36 questionnaire (SF-36)

IPD SHARING:
Plan to Share IPD: No